CLINICAL TRIAL: NCT01717885
Title: Antimalarial Pharmacology in HIV Infected and Uninfected Children and Pregnant Women in Uganda
Brief Title: Antimalarial Pharmacology in Children and Pregnant Women in Uganda
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-04798; R01HD068174 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Malaria; HIV
Keywords: Pharmacokinetics; Antimalarial; HIV; Antiretrovirals; Childhood development; Pregnancy
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples are for drug level measurements,parasite density. RNA samples are for host transcriptional and molecular markers of resistance. Samples are also retained for future use including possible genetic testing for drug metabolism variants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- HIV+children on LPV/r: HIV+ children who are stabilized on a LPV/r based ART regimen
- HIV+ children on nevirapine: HIV+ children who are stabilized on an nevirapine based ART regimen
- HIV+ children on efavirenz: HIV+ children who are stabilized on an efavirenz based ART regimen
- HIV+ pregnant women on LPV/r: HIV+ pregnant women who are stabilized on an LPV/r based ART regimen
- HIV+ pregnant women on NVP: HIV+ pregnant women who are stabilized on an nevirapine based ART regimen
- HIV+ pregnant women on EFV: HIV+ pregnant women stabilized on an efavirenz based ART regimen
- HIV negative children: HIV negative children that will serve as a control for HIV positive children on either a LPV/r, NVP or EFV based ART regimen and will be compared to HIV negative non-pregnant adults
- HIV negative adults: HIV negative adults that will serve as a control for comparing results to HIV negative children and HIV negative pregnant women
- HIV negative pregnant women: HIV negative pregnant women who will serve as a control for HIV positive pregnant women on either a LPV/r, NVP or EFV based ART regimen and will be compared to HIV negative non-pregnant adults

SUMMARY:
The burden of malaria is greatest in children and pregnant women in sub-Saharan Africa. Malaria is one of the most important infectious diseases in the world. Uganda reports among the highest transmission intensities in the world. Children and pregnant women are the most vulnerable populations. HIV is also reported at high rates for these populations. If malaria and HIV require treatment at the same time, there is a high risk for drug-drug interactions. This study will:

1. Determine if the use of anti-HIV medications including lopinavir/ritonavir (LPV/r), nevirapine (NVP) and efavirenz (EFV) will affect the pharmacokinetic (PK) exposure of antimalarial medications (specifically artemether-lumefantrine, AL) during the treatment for uncomplicated malaria in HIV-infected children and pregnant women, and
2. Evaluate the impact of age and pregnancy on the PK exposure of AL.

DETAILED DESCRIPTION:
This study is designed to directly address antimalarial PK and pharmacodynamics (PD) objectives in children and pregnant women, the populations most vulnerable to malaria. This study will focus on the pharmacology of artemether-lumefantrine (AL), the most commonly prescribed anti-malarial drug in sub-Saharan Africa and inform specific dosing guidelines for AL treatment of uncomplicated malaria for these populations. Traditionally, studies have focused on non-pregnant adults, largely ignoring the effects of childhood maturation and pregnancy on drug disposition. This gap in research is specified as a top priority by the WorldWide Antimalarial Resistance Network (WWARN), who emphasize the importance of proper PK and PD study in relevant populations to reduce the threat of ACT drug resistance and treatment failure. This study will allow optimization of ACT regimens, especially in the setting of HIV co-infection and inform use of ART, specifically for the nucleoside analogues, in the setting of malaria and ACT, with the goal of reducing toxicity.

This study complements ongoing PROMOTE trials and provides valuable PK and PD data leveraged to the existing trials, greatly decreasing research costs. This study involves co-enrollment of HIV-infected children and pregnant women already enrolled in PROMOTE which is investigating PI- vs NNRTI-based ART treatment strategies for reducing malaria-related morbidity in HIV and malaria co-infected children and pregnant women. PROMOTE trials were designed in collaboration with Ugandan health care experts and officials and results are expected to rapidly impact Ugandan health policy. This study builds on knowledge gained through PROMOTE. The study also permits enrollment of HIV infected children and pregnant women not in PROMOTE but managed through TDH or other referral site in the Tororo area. Lastly this study will enroll HIV uninfected children, pregnant women and non-pregnant adults.

This study utilizes state-of-the-art PK designs and drug assay methods relying on a combination of intensive and population models to optimize PK/PD analysis. Intensive studies using serial sampling in a relatively small number of subjects will address focused questions on PK exposure while population studies using less frequent sampling in large numbers of subjects will study relationships between PK exposure, clinical response (treatment failure, new infection, and placental malaria), and toxicity (neutropenia) while considering multiple potential covariates. This study includes development and utilization of small volume assay methods for ACT and ART to optimize PK/PD study in children and pregnant women and will be a useful tool for future research trials in resource limited settings.

Rationale for this study is summarized below:

* Dosing guidelines for children and pregnant women have relied on studies carried out in non-pregnant adults
* Children and pregnant women exhibit distinct physiological characteristics that impact how drugs are handled by the body and thus are likely treated improperly
* This gap in research has been deemed an area of high priority by WWARN • Improper dosing may compromise care of acute infection but more importantly contribute to develop of resistance
* ACT therapies must be protected from factors contributing to resistance
* Drug-drug interactions between anti-malarial treatment and ART must be evaluated to assure optimized dosing.
* Drug toxicity, in particular neutropenia, in the setting of HIV-malaria co-infection may be due to important drug-drug interactions
* Intensive PK design resulting in determination of a precise area under the concentration versus time curve (AUC) will permit robust comparisons so that results will inform treatment guidelines and policy for HIV-infected children and pregnant women.
* Once optimized dosing is determined, the PK of this new dosing will be confirmed through follow-up (F/U) studies
* We need state of the art analytical tools to quantitate key drugs in small volume samples collected from vulnerable populations including young children

ELIGIBILITY:
Inclusion Criteria:

ALL PARTICIPANTS

1. Residency within 60 km of the study clinic
2. Agreement to come to clinic for all follow-up clinical and PK evaluations
3. Provision of informed consent

HIV-INFECTED PARTICIPANTS

Children:

1) Enrollment in Promote I or meets enrollment criteria and recruited from TDH/TASO or other referral site

1. 6 months to 8 years of age
2. Weight ≥6 kg
3. Confirmed HIV infection (positive rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
4. On a stable ART regimen for at least 10 days prior to enrollment
5. If co-enrolled from PROMOTE, willingness to undergo intensive PK sampling during a single episode of uncomplicated malaria, and/or population PK/parasite clearance time studies during multiple episodes of uncomplicated malaria.
6. If enrolled from TDH, willingness to undergo intensive PK sampling during a single episode of malaria or population PK/parasite clearance time studies during episodes of uncomplicated malaria.

Pregnant women

1. Enrollment in Promote Project 2 or meets enrollment criteria and recruited from TDH/TASO or other referral site
2. On a stable ART regimen for at least 10 days prior to enrollment
3. Presentation with uncomplicated malaria at the time of enrollment
4. Confirmed pregnancy (apparent pregnancy, positive pregnancy test or pregnancy by ultrasound)
5. Confirmed HIV infection (positive rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
6. 16 years of age or older
7. Estimated gestational age between 12 and 38 weeks by last menstrual period and report of quickening
8. Willingness to undergo intensive PK sampling during episodes of uncomplicated malaria during pregnancy.

HIV UNINFECTED PARTICIPANTS

Children:

1. Enrollment from TDH or other referral site
2. 6 months to 8 years of age
3. Weight ≥6 kg
4. Confirmed HIV negative test (negative rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
5. Presentation with uncomplicated falciparum malaria as indicated by positive smear for malaria parasites along with clinical evidence of infection (fever or history of fever in the past 24 hours) with planned treatment with AL.

7) Willingness to undergo intensive PK sampling during a single episode of malaria or population PK/parasite clearance time studies during episodes of uncomplicated malaria.

Non-pregnant adults:

1. Age ≥ 16 years
2. Confirmed HIV negative test (negative rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment).
3. Presentation with uncomplicated falciparum malaria as indicated by positive smear for malaria parasites along with clinical evidence of infection (fever or history of fever in the past 24 hours) with planned treatment with AL.
4. Negative pregnancy test
5. Willingness to undergo intensive PK sampling during treatment for a single episode of uncomplicated malaria

Pregnant women:

1. Age ≥ 16 years
2. Confirmed HIV negative test (negative rapid HIV test to be confirmed by Western Blot or HIV RNA after enrollment)
3. Confirmed pregnancy (apparent pregnancy, positive pregnancy test or pregnancy by ultrasound)
4. Estimated gestational age between 12 and 38 weeks by last menstrual period and report of quickening
5. Presentation with uncomplicated malaria as indicated by positive smear for malaria parasites along with clinical evidence of infection (fever or history of fever in the past 24 hours) with planned treatment with AL.
6. No evidence of imminent delivery or threatened abortion at the time of presentation with malaria.
7. Willingness to undergo intensive PK sampling during episodes of uncomplicated malaria during pregnancy.

Exclusion Criteria:

1. History of significant comorbidities such as malignancy, active tuberculosis or other WHO stage 4 disease
2. Current infection with non-falciparum species
3. Receipt of any medications known to affect cytochrome p450 (CYP450) metabolism (except ART) within 14 days of study enrollment (see 4.2.2)
4. Hemoglobin < 7.0 g/dL
5. Prior treatment for malaria within 14 days of study enrollment (intensive PK study participants only)
6. Signs or evidence of complicated malaria, defined as unarousable coma OR ANY TWO OF THE FOLLOWING SYMPTOMS: Recent febrile convulsions, altered consciousness, lethargy, unable to drink, unable to stand/sit due to weakness, severe anemia (Hb < 5.0 gm/dL), respiratory distress, jaundice

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected and uninfected children and pregnant women residing in Tororo, Uganda and receiving care at local health care facilities including the Tororo District Hospital (TDH), perinatal facilities, HIV clinics and the IDRC research clinic. HIV uninfected children, pregnant women and non-pregnant adults also enrolled through TDH, perinatal facilities or other area clinics. Each participant can enroll at the time they present to one of the clinics with uncomplicated malaria
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measurement is the area under the plasma concentration versus time curve for all drug analytes. | At time of the last dose of a 6 dose regimen and up to 42 days of F/U
  Pharmacokinetic exposure for the antimalarial medication is estimated through sparse or intensive blood sampling around the last dose and for several days following the last dose.

SECONDARY OUTCOMES:
Malaria reinfection (recrudescence or new infection) | From Day 0 to 42 days of F/U when using artemether-lumefantrine for uncomplicated malaria
  The association between PK exposure and malaria reinfection is the main secondary outcome.
Parasite clearance rate | Days 0 to 42 of follow-up
  To assess the relationship between artemisinin exposure and parasite clearance
AL and ART toxicity | Days 0 to 42 of follow-up
  To assess the relationship between artemether, lumefantrine and antiretroviral exposure and toxicity, particularly neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Francesca T Aweeka, Pharm.D., Study Director — University of California, San Francisco; Sunil Parikh, MD MPH, Principal Investigator — Yale University; Norah Mwebaza, MBChB, MSc, Principal Investigator — Makerere University; Myaing Nyunt, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- IDRC- Tororo Research Clinic and Tororo District Hospital, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nyunt MM, Nguyen VK, Kajubi R, Huang L, Ssebuliba J, Kiconco S, Mwima MW, Achan J, Aweeka F, Parikh S, Mwebaza N. Artemether-Lumefantrine Pharmacokinetics and Clinical Response Are Minimally Altered in Pregnant Ugandan Women Treated for Uncomplicated Falciparum Malaria. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1274-82. doi: 10.1128/AAC.01605-15. PMID 26666942
- [Result] Parikh S, Kajubi R, Huang L, Ssebuliba J, Kiconco S, Gao Q, Li F, Were M, Kakuru A, Achan J, Mwebaza N, Aweeka FT. Antiretroviral Choice for HIV Impacts Antimalarial Exposure and Treatment Outcomes in Ugandan Children. Clin Infect Dis. 2016 Aug 1;63(3):414-22. doi: 10.1093/cid/ciw291. Epub 2016 May 3. PMID 27143666
- [Result] Kajubi R, Huang L, Were M, Kiconco S, Li F, Marzan F, Gingrich D, Nyunt MM, Ssebuliba J, Mwebaza N, Aweeka FT, Parikh S. Parasite Clearance and Artemether Pharmacokinetics Parameters Over the Course of Artemether-Lumefantrine Treatment for Malaria in Human Immunodeficiency Virus (HIV)-Infected and HIV-Uninfected Ugandan Children. Open Forum Infect Dis. 2016 Dec 15;3(4):ofw217. doi: 10.1093/ofid/ofw217. eCollection 2016 Oct. PMID 28018925
- [Derived] Lehane A, Were M, Wade M, Hamadu M, Cahill M, Kiconco S, Kajubi R, Aweeka F, Mwebaza N, Li F, Parikh S. Comparison on simultaneous caillary and venous parasite density and genotyping results from children and adults with uncomplicated malaria: a prospective observational study in Uganda. BMC Infect Dis. 2019 Jun 26;19(1):559. doi: 10.1186/s12879-019-4174-1. PMID 31242863